CLINICAL TRIAL: NCT04911231
Title: Validating Digital Mobility Assessment Using Wearable Technology - the Mobilide-D Clinical Validation Study
Brief Title: Clinical Validation of a Mobility Monitor to Measure and Predict Health Outcomes
Acronym: MOBILISE-D
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0700
Record Dates: First submitted 2021-05-06; First posted 2021-06-02 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background and study aims The ability to move is important for general well-being. Ageing and chronic health conditions can lead to a loss of mobility and a loss of independence. In order to treat mobility loss, tools are needed that can detect and accurately measure mobility. Existing measures of mobility (based on self-reporting and one-off tests) are highly limited. Wearable digital technology (a small device worn on the body) that can be used in the home and the community can provide a simple, accurate and low-cost measure of mobility. The researchers have validated a wearable mobility monitor which can accurately measure how well a person walks by measuring aspects of mobility such as speed and symmetry. The aim of this study is to investigate the ability of the mobility monitor to measure and predict outcomes in proximal femoral fracture (PFF) patients. The digital assessment of mobility developed in this study will be used in clinical trials and in clinical practice.

DETAILED DESCRIPTION:
The study plans to include patients in two groups, both acute (during hospital stay after hip fracture) and subacute (up to 6 months post hip fracture from waiting lists). With this strategy, it is possible to have the life-course of PFF (first 12 months and the time after). Acute phase inclusion is defined as inclusion start on first days after surgery and will be completed within the first 14 days. Subacute phase inclusion is defined as inclusion from waiting lists, where baseline will be conducted up to 6 months after hip fracture surgery.

Fear of falling will be tested using a single question during the acute phase and the short form of the fall efficacy scale international (Short FES-I) for all other assessments. For the acute recruited group of patients (2/3 of included participants), sensor recordings will be made on patients from hospital stay (attached on day 2 after surgery) and continue after discharge (until day 9 depending on battery capacity of the sensors) to be able to monitor and describe DMOs from about 2 days during hospital stay and several days after discharge to be able to evaluate improvement during the acute rehabilitation process. For all other assessments, sensor recordings will be collected for a minimum of 7 full continuous days in line with the core data collection manual.

Hip fracture patients will be tested for sarcopenia according to the updated definitions of the European and US-American working groups. In centers where bioimpedance measurements are possible, participants will receive this measurement as part of the core data collection.

ELIGIBILITY:
Inclusion Criteria:

* Aged 45 or over
* Surgical treatment (fixation or arthroplasty) for a low-energy fracture of the proximal femur (ICD-10 diagnosis S72.0, S72.1, S72.2) as diagnosed on X-rays of the hip and pelvis. Between 3 days and 52 weeks post-surgery
* be able to walk 4 meters

  -.be available for 24 months following the fracture,
* be able to read and understand the briefing note and complete questionnaires feedback
* express their will and sign a consent to participate in follow-up testing, and to wear the motion sensor
* The patient must be a member or beneficiary of a health insurance plan

Exclusion Criteria:

Occurrence of one of the following events in the 3 months preceding the consent enlightened

1. subject with a history of myocardial infarction,
2. Subject hospitalized for unstable angina,
3. Subject with a history of stroke,
4. Subject with a history of coronary bypass surgery (PAC),
5. Subject having had percutaneous coronary intervention (PCI),
6. Subject having had a cardiac resynchronization therapy device implanted (CRTD),

   - Other criteria for non-inclusions
7. Subject with active treatment for cancer or other malignant disease,
8. Subject with uncontrolled congestive heart disease (NYHA class> 3),
9. Subject with acute psychosis or major psychiatric disorders
10. Subject with continued drug addiction.
11. Subject unable to walk prior to hip fracture treatment.
12. The patient is participating in another interventional category I study,
13. l All categories of persons particularly protected under the law French (adults under guardianship, guardianship or safeguard of justice…. articles L1121-8 - L1121-5 - L1121-6 - L1121-7 - L1121-9 of the Health Code Public)

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators will recruit two groups, both acute (during hospital stay after hip fracture) and subacute (up to 6 months post hip fracture from waiting lists). With this strategy the investigators will not only have one segment of the disease, but the life-course of PFF (first 12 months and the time after). Acute phase inclusion is defined as inclusion start on first days after surgery and will be completed within the first 14 days. Subacute phase inclusion is defined as inclusion from waiting lists, where baseline will be conducted up to 6 months after hip fracture surgery.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2024-03-04 (Actual); Study Completion 2024-03-04 (Actual)

PRIMARY OUTCOMES:
Change in the functional component score of the Late-Life Functional Disability Index (LLFDI), that goes from 0 to 100, during 24 months follow-up. | 24 months
  Measured at baseline, 6, 12, 18 and 24 months
Admission to a care home | 6 months
  Assessed from patient records at 6 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Hubert Blain, PD PH, Principal Investigator — University Hospital, Montpellier
Locations (2):
- France (2):
  - Polyclinique Saint-Roch, Montpellier
  - Centre Hospitalier Universitaire de Montpellier, Montpellier